CLINICAL TRIAL: NCT06161116
Title: A Phase 2a, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of MK-6194 in Adult Participants With Systemic Lupus Erythematosus
Brief Title: Efficacy And Safety Of MK-6194 In Adult Participants With Systemic Lupus Erythematosus (MK-6194-006)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6194-006; MK-6194-006 (Other: MSD); 2023-505520-61-00 (Registry Identifier: EU CT); U1111-1291-8716 (Registry Identifier: UTN); jRCT2041230137 (Registry Identifier: jRCT)
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Base Study: Dose 1 (Experimental): Participants receive subcutaneous (SC) MK-6194 dose regimen 1.
  Interventions: Biological: MK-6194
- Base Study: Dose 2 (Experimental): Participants receive SC MK-6194 dose regimen 2.
  Interventions: Biological: MK-6194
- Base Study: Placebo (Placebo Comparator): Participants receive an SC placebo regimen.
  Interventions: Biological: Placebo
- Extension: Dose 1 (Experimental): Participants receive SC MK-6194 dose regimen 1. Participants from the arms "Base Study: Dose 1" or "Base Study: Placebo" may be enrolled in this arm after completing participation in their original arm.
  Interventions: Biological: MK-6194; Biological: Placebo
- Extension: Dose 2 (Experimental): Participants receive SC MK-6194 regimen 2. Participants from the arms "Base Study: Dose 2" or "Base Study: Placebo" may be enrolled in this arm after completing participation in their original arm.
  Interventions: Biological: MK-6194; Biological: Placebo

INTERVENTIONS:
Biological: MK-6194 — SC Injection
  Arms: Base Study: Dose 1; Base Study: Dose 2; Extension: Dose 1; Extension: Dose 2
Biological: Placebo — SC Injection
  Arms: Base Study: Placebo; Extension: Dose 1; Extension: Dose 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of MK-6194 in adult participants with Systemic Lupus Erythematosus. The primary hypothesis is that at least 1 of the MK-6194 arms is superior to placebo in the primary endpoint of percentage of participants with systemic lupus erythematosus responder index (SRI-4) response at Week 28.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of systemic lupus erythematosus (SLE) ≥6 months prior to Screening.
* Is taking at least 1 background therapy (1 immunosuppressant or dapsone and/or 1 antimalarial and/or oral corticosteroids) for SLE.
* Has + antinuclear antibody (+ANA) (titer ≥1:80) or positive anti-double-strand deoxyribonucleic acid (dsDNA) antibody or positive anti-Sm antibody, or positive anti-SSA/Ro antibody.
* Has the presence of at least one of the following manifestations of SLE: Active lupus rash with CLASI-A erythema and scale/hypertrophy combined score >2, or >2 tender and swollen joints in wrists, metacarpophalangeals (MCPs), or proximal interphalangeals (PIPs).
* Has a hybrid Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) total score of ≥6 and clinical hybrid SLEDAI score of ≥4.

Exclusion Criteria:

* Has a concurrent clinically significant disease or clinically relevant laboratory abnormalities, or a history of any illness or medical condition that, in the opinion of the investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
* Has symptomatic heart failure (New York Heart Association class III or IV) or myocardial infarction or unstable angina pectoris within 6 months prior to Screening.
* Has a severe chronic pulmonary disease requiring oxygen therapy.
* Has a transplanted organ which requires continued immunosuppression.
* Has a known systemic hypersensitivity to IL-2, or modified IL-2 including MK-6194, or its inactive ingredients.
* Has a known history of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy and/or splenomegaly.
* Has drug-induced cutaneous lupus erythematosus (CLE) and/or drug-induced SLE in the setting of continued treatment with a causative agent.
* Has active or unstable neuropsychiatric lupus including but not limited to the following: seizure, new or worsening impaired level of consciousness, psychosis, delirium or confused state, aseptic meningitis, cranial neuropathy, cerebrovascular accident, ascending or transverse myelitis, chorea, cerebellar ataxia, mononeuritis multiplex, or demyelinating syndromes.
* Has a diagnosis of Antiphospholipid Syndrome with history of vascular thrombosis, catastrophic APS, or pregnancy morbidity within 6 months prior to Screening.
* Has a history of any malignancy, except for successfully treated non-melanoma skin cancer or localized carcinoma in situ of the cervix.
* Has an active or clinically significant infection requiring hospitalization or treatment with anti-infectives.
* Has evidence of active tuberculosis (TB), latent TB, or inadequately treated TB.
* Has confirmed or suspected COVID-19 infection.
* Has had major surgery within 3 months prior to Screening or has a major surgery planned during the study.
* Is taking more than 1 immunosuppressant.
* Is taking more than 1 oral NSAID (excluding low-dose aspirin [<350 mg/day]) or is taking daily oral nonsteroidal anti-inflammatory drug (NSAID) at greater than the maximum recommended dosage.
* Is currently on any chronic systemic (oral or IV) anti-infective therapy for chronic active infection (such as pneumocystis, cytomegalovirus, herpes zoster, or atypical mycobacteria).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Systemic Lupus Erythematosus Responder Index (SRI-4) Response at Week 28 | Week 28
  The SRI is a composite index used to assess clinical improvement in participants with Systemic Lupus Erythematosus (SLE). The SRI-4 response evaluates global improvement, any significant worsening in unaffected organ systems, and improvements in disease activity, without compromise to the patient's overall condition. SRI-4 response is binary and is either achieved or not achieved by the participant, thus there is no associated score.
Percentage of Participants Experiencing Adverse Events (AEs) | Up to approximately 28 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of Participants Discontinuing Study Treatment Due to an AE | Up to approximately 28 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Percentage of Participants Achieving British Isles Lupus Assessment Group (BILAG)-based Composite Lupus Assessment Response (BICLA) at Week 28 | Week 28
  The BICLA response is a composite global measure of SLE disease activity. It distinguishes between partial and complete improvement in all body systems. BICLA response is binary and is either achieved or not achieved by the participant, thus there is no associated score.
Percentage of Participants Achieving SRI-4 Response at Week 52 | Week 52
  The SRI is a composite index used to assess clinical improvement in patients with Systemic Lupus Erythematosus (SLE). The SRI-4 response evaluates global improvement, any significant worsening in unaffected organ systems, and improvements in disease activity, without compromise to the patient's overall condition. SRI-4 response is binary and is either achieved or not achieved by the participant, thus there is no associated score.
Percentage of Participants Achieving BICLA at Week 52 | Week 52
  The BICLA response is a composite global measure of SLE disease activity. It distinguishes between partial and complete improvement in all body systems. BICLA response is binary and is either achieved or not achieved by the participant, thus there is no associated score.
Percentage of Participants with a Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI)-50 Response at Week 28 | Week 28
  The CLASI-A score is used to evaluate lupus skin manifestations. CLASI-A scores of 0 to 9, 10 to 20, and 21 to 70 represent disease severity of mild, moderate, and severe, respectively. CLASI-50 is 50% of improvement from baseline in the CLASI-A score.
Percentage of Participants with a CLASI-50 Response at Week 52 | Week 52
  The CLASI-A score is used to evaluate lupus skin manifestations. CLASI-A scores of 0 to 9, 10 to 20, and 21 to 70 represent disease severity of mild, moderate, and severe, respectively. CLASI-50 is 50% of improvement from baseline in the CLASI-A score.
Change From Baseline of 28 Joint Count at Week 28 | Baseline and Week 28
  The joint count score is an evaluation of 28 joints in which joints are assessed for presence or absence of swelling and presence or absence of tenderness. The number of affected joints may range from 0 to 28; with higher values corresponding to higher disease activity and lower values to better.
Change From Baseline of 28 Joint Count at Week 52 | Baseline and Week 52
  The joint count score is an evaluation of 28 joints in which joints are assessed for presence or absence of swelling and presence or absence of tenderness. The number of affected joints may range from 0 to 28; with higher values corresponding to higher disease activity and lower values to better.
Change From Baseline of Corticosteroid Dose at Week 28 | Baseline and Week 28
  Participants are assessed for corticosteroid dose change.
Change From Baseline of Corticosteroid Dose at Week 52 | Baseline and Week 52
  Participants are assessed for corticosteroid dose change.
Cumulative Oral Corticosteroid Use Between Week 0 to Week 28 | Up to approximately 28 weeks
  Participants are assessed for total corticosteroid use.
Cumulative Oral Corticosteroid Use Between Week 0 to Week 52 | Up to approximately 52 weeks
  Participants are assessed for total corticosteroid use.
Percentage of Participants Who Achieve Low Level of Disease Activity (LLDAS) at Week 28 | Week 28
  LLDAS is a low disease activity state associated with significant protection against flares and organ damage accrual. It includes both the measurement of disease activity and maintenance of immunosuppressive medications. LLDAS response is binary and is either achieved or not achieved by the participant, thus there is no associated score.
Percentage of Participants Who Achieve LLDAS at Week 52 | Week 52
  LLDAS is a low disease activity state associated with significant protection against flares and organ damage accrual. It includes both the measurement of disease activity and maintenance of immunosuppressive medications. LLDAS response is binary and is either achieved or not achieved by the participant, thus there is no associated score.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (127):
- United States (19):
  - Medvin Clinical Research - Metyas ( Site 0128), Covina, California
  - UCSD - Altman Clinical and Translational Research Institute (ACTRI)-Center for Innovative Therapy ( Site 0110), La Jolla, California
  - Arthritis & Osteoporosis Medical Center - La Palma ( Site 0108), La Palma, California
  - Medvin Clinical Research - Tujunga ( Site 0127), Tujunga, California
  - Denver Arthritis Clinic ( Site 0102), Denver, Colorado
  - Clinical Research of West Florida, Inc. (Clearwater) ( Site 0111), Clearwater, Florida
  - IRIS Research and Development, LLC-Research ( Site 0117), Plantation, Florida
  - Clinical Research of West Florida, Inc ( Site 0124), Tampa, Florida
  - Morehouse School of Medicine ( Site 0146), Atlanta, Georgia
  - Accurate Clinical Research, Inc ( Site 0135), Lake Charles, Louisiana
  - AA Medical Research Center ( Site 0136), Grand Blanc, Michigan
  - Javara - Tryon Medical Partners ( Site 0121), Charlotte, North Carolina
  - DJL Clinical Research, PLLC ( Site 0103), Charlotte, North Carolina
  - University of Oklahoma Health Science Center ( Site 0130), Oklahoma City, Oklahoma
  - Shelby Research, LLC ( Site 0142), Memphis, Tennessee
  - Accurate Clinical Management, LLC. ( Site 0134), Baytown, Texas
  - Epic Medical Research ( Site 0113), DeSoto, Texas
  - Accurate Clinical Research, Inc. ( Site 0133), Houston, Texas
  - SouthWest Rheumatology Research, LLC ( Site 0115), Mesquite, Texas
- Argentina (5):
  - Centro de Investigaciones Médicas Mar del Plata ( Site 0210), Mar del Plata, Buenos Aires
  - Sanatorio Parque ( Site 0205), Rosario, Santa Fe Province
  - Clínica de Nefrología, Urología y Enfermedades Cardiovasculares ( Site 0206), Santa Fe, Santa Fe Province
  - Centro de Investigaciones Médicas Tucuman ( Site 0203), SAN M. de Tucuman, Tucumán Province
  - Instituto de Reumatología ( Site 0201), Mendoza
- Brazil (5):
  - IPC - MT Instituto de Pesquisas Clínicas do Mato Grosso ( Site 0313), Cuiabá, Mato Grosso
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul ( Site 0309), Porto Alegre, Rio Grande do Sul
  - LMK Serviços Médicos S/S-Reumacenter ( Site 0303), Porto Alegre, Rio Grande do Sul
  - Centro Multidisciplinar de Estudos Clinicos ( Site 0302), São Bernardo do Campo, São Paulo
  - Hospital de Base de São José do Rio Preto-CIP - Centro Integrado de Pesquisas ( Site 0311), São José do Rio Preto, São Paulo
- Diex Recherche Sherbrooke ( Site 0003), Sherbrooke, Quebec, Canada
- Chile (6):
  - IC La Serena Research ( Site 0414), La Serena, Coquimbo Region
  - Clinica Dermacross ( Site 0416), Santiago, Region M. de Santiago
  - Complejo Asistencial Dr. Sotero del Rio ( Site 0402), Santiago, Region M. de Santiago
  - CECIM ( Site 0405), Santiago, Region M. de Santiago
  - Centro Internacional de Estudios Clinicos (CIEC) ( Site 0410), Santiago, Region M. de Santiago
  - James Lind Centro de Investigacion del Cancer ( Site 0407), Temuco, Región de la Araucanía
- China (20):
  - The First Afflilated Hospital of Bengbu Medical College-Urology Surgery ( Site 2019), Bengbu, Anhui
  - Anhui Provincial Hospital ( Site 2043), Hefei, Anhui
  - Beijing Peking Union Medical College Hospital-Department of Rheumatology and Immunology ( Site 2001), Beijing, Beijing Municipality
  - Gansu Provincial Hospital ( Site 2065), Lanzhou, Gansu
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University ( Site 2036), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital ( Site 2037), Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University ( Site 2051), Guiyang, Guizhou
  - The Second Afilliated Hospital of Hebei Medical University-Immunology And Rheumatology ( Site 2064), Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of Science &Technology ( Site 2041), Luoyang, Henan
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 2042), Wuhan, Hubei
  - The First Affiliated Hospital of Nanhua University ( Site 2061), Hengyang, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Te ( Site 2006), Baotou, Inner Mongolia
  - Affiliated Hospital of Nantong University ( Site 2027), Nantong, Jiangsu
  - Pingxiang People's Hospital ( Site 2005), Pingxiang, Jiangxi
  - Jilin Province People's Hospital ( Site 2033), Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University ( Site 2056), Xi'an, Shaanxi
  - Renji Hospital Shanghai Jiao Tong University School of Medicine ( Site 2053), Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital ( Site 2029), Taiyuan, Shanxi
  - The First Affiliated Hospital Of Chengdu Medical College ( Site 2052), Chengdu, Sichuan
  - Tianjin Medical University General Hospital-Rheumatism and Immunology ( Site 2011), Tianjin, Tianjin Municipality
- Colombia (7):
  - Salud SURA Industriales ( Site 0508), Medellín, Antioquia
  - Centro Integral de Reumatología del Caribe ( Site 0501), Barranquilla, Atlántico
  - Clinica de la Costa S.A.S. ( Site 0502), Barranquilla, Atlántico
  - Preventive Care ( Site 0507), Chía, Cundinamarca
  - Healthy Medical Center S.A.S ( Site 0505), Zipaquirá, Cundinamarca
  - Fundación Valle del Lili ( Site 0506), Cali, Valle del Cauca Department
  - Centro de Estudios de Reumatología y Dermatología SAS ( Site 0512), Cali, Valle del Cauca Department
- France (6):
  - CHU Bordeaux Haut-Leveque ( Site 1007), Pessac, Aquitaine
  - Centre Hospitalier Saint Joseph - Saint Luc ( Site 1003), Lyon, Auvergne-Rhône-Alpes
  - CHU Rangueil ( Site 1008), Toulouse, Haute-Garonne
  - CHU Montpellier Lapeyronie Hospital-Rhumatologie ( Site 1006), Montpellier, Herault
  - Hopital Claude Huriez - CHU de Lille ( Site 1005), Lille, Nord
  - Centre Hospitalier Universitaire de Saint Étienne - Hôpital Nord ( Site 1009), Saint Priest En Jarez, Pays de la Loire Region
- Guatemala (3):
  - Clínica Médica Especializada en Pediatría e Infectología Pediátrica - Dr. Mario Melgar ( Site 0602), Guatemala City
  - CELAN,S.A ( Site 0603), Guatemala City
  - Clinica Medica Especializada en Medicina Interna y Reumatología ( Site 0601), Guatemala City
- Italy (7):
  - Istituto Clinico Humanitas Research Hospital ( Site 1310), Rozzano, Milano
  - Fondazione Policlinico Universitario Campus Bio-Medico ( Site 1307), Rome, Roma
  - Azienda Ospedaliero Universitaria Senese-Medicina Interna e Specialistica ( Site 1306), Siena, Tuscany
  - Azienda Ospedale - Università Padova-Department of Medicine-DIMED ( Site 1309), Padua, Veneto
  - AOU Careggi ( Site 1311), Florence
  - Azienda Ospedaliera Universitaria dell'Università "Luigi Van-UNITA'OPERATIVA DI REUMATOLOGIA, DIPAR ( Site 1305), Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -UOC Reumatologia ( Site 1304), Roma
- Japan (12):
  - Japan Community Healthcare Organization Chukyo Hospital ( Site 2107), Nagoya, Aichi-ken
  - St. Marianna University Hospital ( Site 2121), Kawasaki, Kanagawa
  - Tohoku University Hospital ( Site 2116), Sendai, Miyagi
  - Yuuai Medical Center ( Site 2122), Tomigusuku, Okinawa
  - Shimane University Hospital ( Site 2119), Izumo, Shimane
  - Dokkyo Medical University Hospital ( Site 2118), Shimotsuga, Tochigi
  - Nihon University Itabashi Hospital ( Site 2105), Itabashiku, Tokyo
  - Showa Medical University East Hospital ( Site 2123), Shinagawa, Tokyo
  - Chiba University Hospital ( Site 2120), Chiba
  - NHO Chiba Medical Center Chibahigashi National Hospital ( Site 2112), Chiba
  - Okayama University Hospital ( Site 2106), Okayama
  - Osaka Keisatsu Hospital ( Site 2117), Osaka
- Malaysia (4):
  - Hospital Canselor Tuanku Muhriz UKM ( Site 2225), Cheras, Kuala Lumpur
  - University Malaya Medical Centre-Clinical Investigation Centre (CIC) ( Site 2222), Lembah Pantai, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan-Medical Outpatient Department ( Site 2224), Kuantan, Pahang
  - Hospital Taiping ( Site 2221), Taiping, Perak
- Mexico (12):
  - Morales Vargas Centro de Investigacion ( Site 0710), León, Guanajuato
  - Centro Integral en Reumatologia ( Site 0701), Guadalajara, Jalisco
  - Centro de Atención en Enfermedades Inflamatorias CATEI ( Site 0707), Guadalajara, Jalisco
  - Clinica de Investigacion en Reumatologia y Obesidad S. C. ( Site 0705), Guadalajara, Jalisco
  - Centro de Estudios de Investigacion Basica y Clinica ( Site 0708), Guadalajara, Jalisco
  - RM Pharma Specialists ( Site 0711), Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran ( Site 0713), Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Rheumatology ( Site 0706), Monterrey, Nuevo León
  - Centro Potosino de Investigación Médica ( Site 0703), San Luis Potosí City, San Luis Potosí
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion Clinica en Yucatan ( Site 0712), Mérida, Yucatán
  - ICARO Investigaciones en Medicina ( Site 0702), Chihuahua City
  - Clinstile, S.A. de C.V. ( Site 0709), Distrito Federal
- Philippines (3):
  - Mary Mediatrix Medical Center ( Site 2303), Lipa City, Batangas
  - ST. LUKE'S MEDICAL CENTER ( Site 2304), Quezon City, National Capital Region
  - Iloilo Doctors' Hospital ( Site 2301), Iloilo City
- Poland (8):
  - Medyczne Centrum Hetmańska ( Site 1406), Poznan, Greater Poland Voivodeship
  - Prywatna Praktyka Lekarska Prof. UM dr hab. med. Pawel Hrycaj ( Site 1402), Poznan, Greater Poland Voivodeship
  - MICS Centrum Medyczne Bydgoszcz ( Site 1410), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Plejady ( Site 1407), Krakow, Lesser Poland Voivodeship
  - Zespół Poradni Specjalistycznych Reumed Filia nr 1 Wallenroda ( Site 1408), Lublin, Lublin Voivodeship
  - MICS Centrum Medyczne Warszawa ( Site 1411), Warsaw, Masovian Voivodeship
  - Nova Reuma Społka Partnerska ( Site 1405), Bialystok, Podlaskie Voivodeship
  - NZOZ BIF-MED ( Site 1409), Bytom, Silesian Voivodeship
- Spain (5):
  - CHUAC-Complejo Hospitalario Universitario A Coruña-Reumatologia ( Site 1604), A Coruña, La Coruna
  - HOSPITAL CLINICO DE VALENCIA ( Site 1608), Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d'Hebron-Rheumatology ( Site 1601), Barcelona
  - Hospital Quiron Infanta Luisa-Unidad de investigacion de Reumatologia ( Site 1602), Seville
  - Hospital Universitario Rio Hortega ( Site 1606), Valladolid
- Turkey (Türkiye) (4):
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi ( Site 1709), Kadıköy, Istanbul
  - ANKARA UNIVERSITY IBNI SINA HOSPITAL-Rheumatology Department ( Site 1703), Ankara
  - Ankara Bilkent Şehir Hastanesi-Rheumatology ( Site 1702), Ankara
  - Sakarya Training and Research Hospital-Rheumatology ( Site 1708), Sakarya

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26196&tenant=MT_MSD_9011